CLINICAL TRIAL: NCT06394635
Title: Investigation of the Effect of Using Plantar Flexion Resistant Ankle-Foot Orthosis in Stroke Patients With Genurecurvatum Gait
Brief Title: Use of Plantar Flexion Resistant Ankle-Foot Orthosis in Stroke Patients With Genurecurvatum Gait
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Other Study IDs: 349c6c25d7a64a22
Record Dates: First submitted 2024-04-28; First posted 2024-05-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Stroke Patients with Genurecurvatum Gait: Stroke patients with genurecurvatum gait will be included.

SUMMARY:
Hypothesis 1:

Ho: Ankle-foot orthosis, which fixes the ankle at different angles (3 degrees dorsiflexion - 5 degrees dorsiflexion), has no effect on knee hyperextension control in stroke patients with genurecurvatum gait.

H1: Ankle-foot orthosis, which fixes the ankle at different angles (3 degrees dorsiflexion - 5 degrees dorsiflexion), has an effect on knee hyperextension control in stroke patients with genurecurvatum gait.

Hypothesis 2:

Ho: Ankle-foot orthosis, which fixes the ankle at different angles (3 degrees dorsiflexion - 5 degrees dorsiflexion), has no effect on pelvic movements in stroke patients with genurecurvatum gait.

H1: Ankle-foot orthosis, which fixes the ankle at different angles (3 degrees dorsiflexion - 5 degrees dorsiflexion), has an effect on pelvic movements in stroke patients with genurecurvatum gait.

DETAILED DESCRIPTION:
Kinematic evaluation of the gaits of stroke patients in 3 different situations will be made in the motion analysis system. Patients will be asked to walk at a normal walking pace for a distance of only 5 meters. Patients will walk the 5-meter distance first without the Ankle-Foot Orthosis, then with the Ankle-Foot Orthosis adjusted at 3 degrees of dorsiflexion, and then with the Ankle-Foot Orthosis adjusted at 5 degrees of dorsiflexion.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months have passed since the stroke incident
* Ambulating with or without a walking aid (walker, cane or tripod)
* Being between 0-3 points according to the Modified Rankin Scoring
* Getting a score of 24 or above from the Mini Mental Test
* Presence of hyperextension in the stance phase of gait
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of more than one stroke
* Known presence of dementia
* Having a known orthopedic, psychiatric or other neurological disease
* There is a situation that prevents communication
* Having a history of surgery involving the lower extremities and gait

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke Patients with Genurecurvatum Gait
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Movement Analysis | Baseline
  Reflective signs will be placed on certain anatomical points on the participants and the participants will be asked to walk at a distance of 5 meters. The three-dimensional positions of these reflective signs will be captured with the 8-camera Vicon motion capture system and recorded on the computer using Blade software.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Korkusuz, PhD, Principal Investigator — Atılım University; Büşra Seçkinoğulları Korkusuz, MSc, Study Chair — Hacettepe University; Ayşenur Özcan, MSc, Study Chair — Çankırı Karatekin University; Ferdi Yavuz, Assoc.Prof., Study Chair — European University of Lefke; Nihat Özgören, PhD, Study Chair — Hacettepe University; Serdar Arıtan, Assisst.Prof, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kobayashi T, Orendurff MS, Singer ML, Gao F, Daly WK, Foreman KB. Reduction of genu recurvatum through adjustment of plantarflexion resistance of an articulated ankle-foot orthosis in individuals post-stroke. Clin Biomech (Bristol). 2016 Jun;35:81-5. doi: 10.1016/j.clinbiomech.2016.04.011. Epub 2016 Apr 23. PMID 27136122
- [Background] Bae DY, Shin JH, Kim JS. Effects of dorsiflexor functional electrical stimulation compared to an ankle/foot orthosis on stroke-related genu recurvatum gait. J Phys Ther Sci. 2019 Nov;31(11):865-868. doi: 10.1589/jpts.31.865. Epub 2019 Nov 26. PMID 31871367
- [Background] Geerars M, Minnaar-van der Feen N, Huisstede BMA. Treatment of knee hyperextension in post-stroke gait. A systematic review. Gait Posture. 2022 Jan;91:137-148. doi: 10.1016/j.gaitpost.2021.08.016. Epub 2021 Aug 24. PMID 34695721